CLINICAL TRIAL: NCT03845868
Title: Tongji-Ezhou Prospectively Cohort Study
Brief Title: Tongji-Ezhou Study
Acronym: TJEZ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Liegang Liu, Vice dean of School of Public Health, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: TJEZ2013
Record Dates: First submitted 2019-02-14; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Diabetes; Cardiovascular Diseases; Obesity; Metabolic Syndrome; Nutritional and Metabolic Diseases; Environmental Exposure; Risk Factor, Cardiovascular
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Obesity; Metabolic Syndrome; Nutritional and Metabolic Diseases | interventions — Diet; Environmental Exposure; Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, and DNA were collected by clinicians during the morning after the examinees. Blood samples (5 ml) are collected with ethylenediamine tetra acetic acid anticoagulant tube from peripheral vessels. Plasma, buffy coat, and red blood cell layer are separated. The samples are stored at -80°C for future analyses. All bio-samples will be tracked through an electronic database.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Egang hospital physical examination center
  Interventions: Other: Dietary and environmental exposure (Observational study)
- Ezhou CDC physical examination center
  Interventions: Other: Dietary and environmental exposure (Observational study)

INTERVENTIONS:
Other: Dietary and environmental exposure (Observational study)

SUMMARY:
Tongji-Ezhou study (TJEZ) is a prospective cohort study launched at 2013 in EZhou city, Hubei province, with the goal of recruiting and assessing 10,000 individuals and then following them for at least 2 decades. In addition, blood samples would be collected every 3-5 years among 6000 of them to investigate the nutritional biomarkers and potential determinants of chronic diseases such as obesity, type 2 diabetes, metabolic syndrome, and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* (i) permanent residence in Ezhou district (minimum of 9 months); (ii) written informed consent; (iii) age ≥ 20 years old at the time of enrolling in the study.

Exclusion Criteria:

* (i) with chemotherapy or radiotherapy for cancer and other severe diseases.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Samples were collected at two medical centrals (retired employees at Egang hospital and working employees at Ezhou CDC). The Retirement Office of Egang hospital and Health checkup center of CDC provided a list of the individuals and invited them to participant in our study.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-04-16 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of diabetes | 5 years
  Type 2 diabetes was diagnosed when FPG ≥ 7.0 mmol/L and/or OGTT2h ≥ 11.1 mmol/L, or using diabetic medication (self-report).
Incidence of metabolic syndrome | 5 years
  Metabolic syndrome is defined as using the updated National Cholesterol Education Program/Adult Treatment Panel III criteria for Asian Americans. These criteria require three or more of the following components: (1) central obesity (waist circumference of ≥90 cm for men or ≥80 cm for women), (2) triglycerides of ≥1.7 mmol/L, (3) HDL-C of <1.03 mmol/L for men or <1.30 mmol/L for women, (4) blood pressure of ≥130/85 mmHg or on medication for hypertension, and (5) fasting glucose of ≥5.6 mmol/L.
Diabetic complications | mean follow up of 10 years
  Development of diabetic complications
Incidence of cardiovascular diseases | mean follow up of 10 years
  Cardiovascular death, stroke, myocardial infarction, heart failure

CONTACTS AND LOCATIONS:
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sun T, Deng Y, Geng X, Fang Q, Li X, Chen L, Zhan M, Li D, Zhu K, Li H, Liu L. Plasma Alkylresorcinol Metabolite, a Biomarker for Whole-Grain Intake, Is Inversely Associated with Risk of Nonalcoholic Fatty Liver Disease in a Case-Control Study of Chinese Adults. J Nutr. 2022 Apr 1;152(4):1052-1058. doi: 10.1093/jn/nxab404. PMID 35091747